CLINICAL TRIAL: NCT07083284
Title: Acute Kidney Injury in Neonatal ICU in Assuit University
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omnia Zakaria Mostafa, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: AKI neonatal ICU
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: patients with Age from 0 to 28 days presented with acute kidney injury on based of raised renal chemistry, An increase in serum creatinine (e.g., >0.3 mg/dL or >50% from baseline) , Oliguria (urine output less than 1 mL/kg/h for more than 6 hours).

SUMMARY:
The kidneys of neonates are particularly susceptible to hypoperfusion because of the physiologic characteristics of neonatal kidneys, including high renal vascular resistance, high plasma renin activity, low glomerular filtration rate (GFR), decreased intracortical perfusion rate, and decreased reabsorption of sodium in proximal convoluted tubules in the first day of neonatal life (1) Acute kidney injury (AKI) occurs commonly in the neonatal intensive care unit (NICU) and is associated with increase morbidity and mortality. Furthermore, those who develop neonatal AKI may be at increased risk for the development of chronic kidney disease (CKD). With ongoing study, the definition of neonatal AKI has evolved and been standardized, improving our ability to quantify and describe the epidemiology and outcomes associated with neonatal AKI (2) Acute kidney injury (AKI) is defined as kidneys' inability to excrete nitrogenous waste products and maintain fluid and electrolyte homeostasis. It is fairly common in newborn population and is a major contributing factor of neonatal mortality and morbidity (3) Acute kidney injury (AKI), frequently involving patients admitted to the neonatal intensive care unit (NICU), is associated with poor outcomes and affects 18-70% of critically ill neonates. Although the real incidence of AKI in neonates is uncertain, with wide and various ranges, due to several definitions and diagnostic methods, more immature and ill neonates are characterized by the highest risk of AKI (4) Patients with congenital heart disease, perinatal asphyxia, premature birth or a low birth weight, and necrotizing enterocolitis, as well as neonates who receive nephrotoxic medications or require extracorporeal life support, represent high-risk populations. According to the Worldwide Acute Kidney Injury Epidemiology in Neonates (AWAKEN) data, one episode of AKI, related to an increased length of hospitalization and mortality rate, was observed in 30% of critically ill neonates (5) To apply personalized therapeutic approaches to AKI, an adequate and early diagnosis could reduce or avoid subclinical and precocious renal injuries and their related effects, requiring chronic follow-up, as suggested by the Clinical Practice Guidelines for Acute Kidney Injury (KDIGO), recommending a nephrological evaluation after three months, if an AKI event occurs (6)

The precocious diagnosis of AKI based on urinary output and serum creatinine (sCr) levels represents one of the hardest challenges in clinical practice. Several biomarkers and clinical scores were assessed to predict neonatal AKI, to identify the stage of injury and not the damage, to anticipate late rises in sCr values and to reveal an already compromised renal function (7)

ELIGIBILITY:
Inclusion Criteria:

* • Age from 0 to 28 days presented with acute kidney injury on based of raised renal chemistry, An increase in serum creatinine (e.g., >0.3 mg/dL or >50% from baseline) , Oliguria (urine output less than 1 mL/kg/h for more than 6 hours).

  * Other biomarkers of kidney injury (e.g., elevated urinary biomarkers such as NGAL, KIM-1) ( if available)
  * Parental consent: Neonates whose parents or legal guardians provide informed consent for participation in the study

Exclusion Criteria:

* • Post-operative neonates.

  * Cases with gross congenital anomalies of the kidney and urinary tract.
  * Neonates with a maternal history of kidney failure.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with Age from 0 to 28 days presented with acute kidney injury on based of raised renal chemistry, An increase in serum creatinine (e.g., >0.3 mg/dL or >50% from baseline) , Oliguria (urine output less than 1 mL/kg/h for more than 6 hours).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
incidance of acute kidney injery | 30 day
  incidance of acute kidney injery of neonate